CLINICAL TRIAL: NCT06817642
Title: Predicting Language Recovery in Acute Stroke Patients in the Neurovascular Intensive Care Unit: An Exploratory Study With the Core Assessment of Language Processing.
Acronym: PREDICT-CALAP
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220542
Record Dates: First submitted 2023-07-05; First posted 2025-02-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-02

CONDITIONS: Stroke Patients
Keywords: Stroke; Aphasia; Language abilities; Cognitive abilities; Prediction of function recovery
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data recovery from language and cognitive assessment — Data recovery from language assessment: Core Assessment of LAnaguage Processing, and from neuropsychological assessment : Montreal Cognitive Assessment, Trail Making Test, Batterie Rapide d'Efficience Frontale (BREF), animal fluency, 5 words of Dubois, Ne

SUMMARY:
Introduction:

Stroke affects one person every 4 minutes in France (i.e. more than 140,000 new cases per year) resulting in cognitive and motor disorders. Aphasia is one of the most devastating cognitive disorders that persist in the late phase. However, early treatment of aphasia can improve the effects of rehabilitation.

Identifying, as early as possible, the patients most at risk of presenting persistent language disorders in the late phase would make it possible to improve their management and increase the effects of cognitive rehabilitation on their language abilities.

The aim of this project is to evaluate whether the Core Assessment of Language Processing (CALAP) assessed in the acute phase of stroke can predict language abilities in the late phase.

Hypothesis/Objective:

The primary objective is to determine whether the language abilities of patients in the acute phase of stroke can be used to predict language abilities in the late phase. Secondary objectives are to determine whether prediction can be improved with (1) brain MRI data and (2) neuropsychological assessment data. The (3) secondary objective is to determine whether cognitive abilities at the chronic phase can be predicted by language performance in the acute phase. The (4) secondary objective is to assess whether language rehabilitation modifies the predictive power of the language abilities assessed with the CALAP.

Method:

Patients will be included during their hospitalization after a brain vascular injury (acute phase, up to 21 days of hospitalization). After discharge, they will return for a post-stroke assessment between 3 and 18 months after the acute phase.

During these two visits, a clinical and neurological examination, a neuropsychological assessment and an MRI will be performed.

A prediction model (development and validation) will be used for all objectives using a linear regression model with cross validation. The entire sample consists of stroke patients.

The study is single-center and will have a total duration of 6 years with an estimated 570 patients included.

Conclusion:

Predicting the language abilities of a post-stroke patient will improve clinical management and direct patients requiring language rehabilitation to appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 18 and 85 years old
* Inpatient in the initial phase of stroke (between 0 and 21 days after stroke)
* Hemispheric stroke, ischemic or haemorrhagic
* Ability to participate in tests
* Francophone
* 4≤ NIHSS score ≤21 or if NIHSS score < 4, LAST score [0-13]
* Non-opposition to participation in tests

Exclusion Criteria:

* Severe alertness impairment incompatible with test participation, NIHSS score 1a. different from 0
* Severe overall intellectual deterioration incompatible with test participation
* Patients who may have a visual or hearing impairment incompatible with participation in CALAP
* History of stroke
* Posterior fossa stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients (hemispheric stroke, ischemic or hemorrhagic).
Sampling Method: Probability Sample
Enrollment: 570 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Language recovery prediction with Core Assessment of Language Processing score | 18 months after stroke
  the objective is to predict from stroke patient's language performance in the acute phase, his or her language performance in the late phase

SECONDARY OUTCOMES:
Improving CALAP recovery prediction using MRI data | 18 months after stroke
  Improvement of the predictive value of the CALAP score in the acute phase using brain MRI data (lesion volume, lesion location, and/or percentage of disconnected fibers measured by MRI).
Improving CALAP recovery prediction using neuropsychological data | 18 months after stroke
  Improvement of the predictive value of the CALAP score in the acute phase using neuropsychological assessment data collected in the acute phase.
Cognitive recovery prediction with Core Assessment of Language Processing score | 18 months after stroke
  The objective is to predict cognitive abilities at the chronic phase based on language performance in the acute phase
Improving CALAP recovery prediction using language rehabilitation data | 18 months after stroke
  The objective is to assess whether language rehabilitation modifies the predictive power of the language abilities assessed with the CALAP

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hôpitaux de Paris - Hôpital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No